CLINICAL TRIAL: NCT07085442
Title: NodeSMART - Audit of Targeted Sentinel Node Biopsy (TSNB) in Patients With Limited Nodal Disease Undergoing Primary Surgery
Brief Title: Audit of Targeted Sentinel Node Biopsy (TSNB) in Patients With Limited Nodal Disease Undergoing Primary Surgery
Acronym: NodeSMART
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Amit Goyal, Chief Investigator, University Hospitals of Derby and Burton NHS Foundation Trust
Other Study IDs: PID 46
Record Dates: First submitted 2025-07-09; First posted 2025-07-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Axillary Lymph Nodes Dissection; Axillary Metastases; Sentinel Lymph Node Biopsy (SLNB); Node Positive Breast Cancer; Axilla; Breast; Axillary Ultrasound
Keywords: Targeted Axillary Dissection; Targeted Sentinel Node Biopsy; NodeSMART; Breast Cancer; Sentinel Node Biopsy; Axillary Lymph Nodes Dissection; Axillary Node Clearance
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with biopsy proven nodal metastases (cN1) and not receiving neoadjuvant chemotherapy: Patients with T1 or T2 tumours with biopsy proven nodal metastases (cN1) and with ≤2 abnormal nodes on axillary ultrasound
  Interventions: Procedure: Targeted Sentinel Node Biopsy (TSNB)

INTERVENTIONS:
Procedure: Targeted Sentinel Node Biopsy (TSNB) — Targeted Sentinel Node Biopsy will be performed according to routine local practice. The procedure has been standardised for the post-NACT setting as part of the ongoing ATNEC trial. Sites are advised to follow the ATNEC protocol in the primary surgery setting, using either a dual- or single-tracer sentinel node biopsy technique, with localisation and removal of the marked biopsy proven positive node, and removal of at least 3 nodes.

SUMMARY:
Axillary ultrasound scan (AUS) is routinely employed in the UK for preoperative axillary staging and can diagnose approximately 50 - 80% of node positive patients when combined with percutaneous needle biopsy techniques (either core-biopsy or fine-needle aspiration cytology). It is recognised that nodal burden is generally higher in clinically node negative patients with abnormal nodes on AUS and confirmed on needle-biopsy to be histologically positive than patients diagnosed as node positive on sentinel node biopsy (SNB). However, up to 40% of biopsy-proven node positive patients are found to have fewer than 3 involved nodes on subsequent axillary lymph node dissection (ALND) and are potential candidates for less extensive axillary surgery with axillary radiotherapy (ART) rather than ALND. The total number of abnormal nodes on ultrasound is a key predictor of overall nodal tumour burden.

The AMAROS and OTOASOR trials randomised patients with up to 2 positive sentinel nodes to either ALND or ART. These trials were conducted around the turn of the millennium and before routine use of AUS and therefore would have included a significant number of patients who were radiologically node positive (cN1). Likewise, the ACOSOG Z0011 trial that randomised a similar group of patients to either ALND or observation only, did not incorporate routine AUS and would have included some (radiological) cN1 patients. These trials revealed no adverse impact on disease-free or overall survival from omission of completion ALND.

Targeted axillary dissection (TAD) was introduced a few years ago to reduce the false negative rate of SNB following neoadjuvant chemotherapy (NACT) and has been standardised as part of the ongoing ATNEC trial [ClinicalTrials.govNCT04109079]. This technique for axillary staging after NACT is increasingly being adopted in the UK and elsewhere. TAD is technically more straightforward and less challenging in patients undergoing primary surgery with no concerns about clip migration consequent to nodal shrinkage as part of treatment response to NACT. Furthermore, the risk of under-treating the axilla is offset by the protocol: if no disease is identified in the targeted nodes (false-negative case), then patients proceed to ALND, thereby ensuring adequate treatment. Unlike TAD following NACT, the presence of viable tumour within the sampled nodes is mandatory and finding fibrosis is irrelevant except as a response to nodal biopsy per se.

Current ASCO guidelines support both SNB and TAD as staging options for patients with ultrasound-detected, biopsy-confirmed nodal disease. The Edinburgh randomised trials comparing four-node sampling with ALND demonstrated significantly lower arm morbidity with node sampling, supporting TAD as a clinically appropriate alternative in this patient population.

The UK-ANZ POSNOC trial randomised 1,900 patients with <3 macrometastases to either no further axillary treatment or additional axillary treatment. The study included cN1 patients with biopsy-confirmed nodal metastases who underwent sentinel node biopsy or TAD. Patients with <3 macrometastases on final histology were randomised to receive no further axillary treatment or proceed with additional axillary treatment (ALND or ART). POSNOC trial will answer whether further axillary treatment provides any benefit in patients with low volume nodal disease on SNB or TAD.

Notably, patients with biopsy-confirmed metastases and <3 macrometastases on SNB/TAD are biologically and clinically similar to patients with normal AUS who are later found to have low-volume disease on SNB. Clinical decision-making and patient outcomes are driven by tumour biology and overall disease burden rather than the method of nodal disease detection. Furthermore, AUS sensitivity is operator dependent and whether FNA or core biopsy was used to sample the node. A patient considered node negative on AUS by one radiologist may be diagnosed with core biopsy confirmed nodal metastases with another radiologist. Pending the results of POSNOC trial, patients with less than 3 macrometastases are generally advised further axillary treatment, and ART is preferred over ALND to reduce the risk of lymphoedema.

NodeSMART is a prospective audit collecting data on patients undergoing TAD in the primary surgery setting. Its goal is to audit surgical outcomes and benchmark them against - a) Comparing technical outcomes with those from sentinel node biopsy in the primary surgery setting and TAD performed after neoadjuvant chemotherapy. b) Assessing rates of arm lymphoedema and disease progression relative to findings from the AMAROS and Z11 trials, and the POSNOC trial once results are available. The term "Targeted Axillary Dissection" is somewhat misleading in this context, as the marked (biopsied) node is removed alongside sentinel nodes - not in isolation. NodeSMART therefore refers to the procedure more accurately as Targeted Sentinel Node Biopsy (TSNB).

DETAILED DESCRIPTION:
Guidelines for node marking:

Sites are advised to follow the same standards used in the ongoing ATNEC breast cancer trial. At least three nodes should be removed to allow adequate assessment of nodal tumour burden.

Timing:

The node may be marked at the time of needle biopsy or at a separate visit.

Technique:

Node may be marked using any technique e.g. clip or coil (with or without skin mark), black dye, magnetic seeds or reflector.

Black dye node marking:

Inject 0.2-0.4 ml of black dye into the cortex of the node Do not inject around the node or into the needle tract

If the marked node is not found or if multiple black nodes are identified the surgeon may stop once a total of four nodes have been removed

Single vs multiple node marking:

It is not necessary to mark more than one node, even if multiple nodes are biopsied or appear malignant. The most abnormal-appearing node should be marked.

ELIGIBILITY:
Inclusion Criteria:

* cT1-2N1M0 breast cancer
* FNA or core biopsy confirmed axillary nodal metastases
* ≤2 abnormal nodes on imaging
* Undergo a dual tracer or single tracer sentinel node biopsy along with removal of the marked node (Targeted Sentinel Node Biopsy, TSNB)
* 1 or 2 macrometastases identified in the removed nodes, with at least three nodes removed
* If the sentinel node(s) cannot be localised on SNB: axillary node sampling should be performed, the patient will be eligible if 1 or 2 macrometastases are identified in the removed nodes, with at least three nodes removed.
* If the node is not marked or the marked node is not removed, the patient will be eligible if 1 or 2 macrometastases are identified in the removed nodes, with at least three nodes removed.

Exclusion Criteria:

* Neoadjuvant chemotherapy
* Previous ipsilateral axillary nodal surgery
* cT3-4 breast cancer
* ≥3 abnormal nodes on imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cT1-2N1M0 breast cancer patients aged 18 years or older, with needle biopsy proven nodal metastases, ≤2 abnormal nodes on imaging, and are undergoing sentinel node biopsy and removal of the marked involved node.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Patients with ≤2 nodal macrometastases identified on histology. | 12 months
  To determine the number of patients with fewer than 3 nodal macrometastases on final histology, and assess whether ultrasound-detected abnormal nodes and tumour characteristics can predict axillary nodal burden.
Patients with ≤2 nodal macrometastases identified on histology. | 24 months
  To determine the number of patients with fewer than 3 nodal macrometastases on final histology, and assess whether ultrasound-detected abnormal nodes and tumour characteristics can predict axillary nodal burden.
Patients with ≤2 nodal macrometastases identified on histology. | 36 months
  To determine the number of patients with fewer than 3 nodal macrometastases on final histology, and assess whether ultrasound-detected abnormal nodes and tumour characteristics can predict axillary nodal burden.
Patients with ≤2 nodal macrometastases identified on histology. | 48 months
  To determine the number of patients with fewer than 3 nodal macrometastases on final histology, and assess whether ultrasound-detected abnormal nodes and tumour characteristics can predict axillary nodal burden.
Patients with ≤2 nodal macrometastases identified on histology. | 60 months
  To determine the number of patients with fewer than 3 nodal macrometastases on final histology, and assess whether ultrasound-detected abnormal nodes and tumour characteristics can predict axillary nodal burden.
Identification rate of marked node | 12 months
  Identification rate of marked biopsied node at axillary surgery
Identification rate of marked node | 24 months
  Identification rate of marked biopsied node at axillary surgery
Identification rate of marked node | 36 months
  Identification rate of marked biopsied node at axillary surgery
Identification rate of marked node | 48 months
  Identification rate of marked biopsied node at axillary surgery
Identification rate of marked node | 60 months
  Identification rate of marked biopsied node at axillary surgery
False negative rate of targeted sentinel node biopsy | 12 months
  False negative rate of targeted sentinel node biopsy (FN/TP+FN)
False negative rate of targeted sentinel node biopsy | 24 months
  False negative rate of targeted sentinel node biopsy (FN/TP+FN)
False negative rate of targeted sentinel node biopsy | 36 months
  False negative rate of targeted sentinel node biopsy (FN/TP+FN)
False negative rate of targeted sentinel node biopsy | 48 months
  False negative rate of targeted sentinel node biopsy (FN/TP+FN)
False negative rate of targeted sentinel node biopsy | 60 months
  False negative rate of targeted sentinel node biopsy (FN/TP+FN)
Arm lymphoedema | 12 months
  Arm lymphoedema self reported by the patient or identified during routine care, resulting in referral to a lymphoedema clinic.
Arm lymphoedema | 24 months
  Arm lymphoedema self reported by the patient or identified during routine care, resulting in referral to a lymphoedema clinic.
Arm lymphoedema | 36 months
  Arm lymphoedema self reported by the patient or identified during routine care, resulting in referral to a lymphoedema clinic.
Arm lymphoedema | 48 months
  Arm lymphoedema self reported by the patient or identified during routine care, resulting in referral to a lymphoedema clinic.
Arm lymphoedema | 60 months
  Arm lymphoedema self reported by the patient or identified during routine care, resulting in referral to a lymphoedema clinic.

SECONDARY OUTCOMES:
Axillary recurrence | 12 months
  Axillary recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence in lymph nodes draining the primary tumour site, i.e. nodes in the ipsilateral axilla, infraclavicular fossa, supraclavicular fossa and interpectoral area. The date of axillary recurrence is the date on which imaging or pathology report (whichever comes first) confirms axillary recurrence.
Axillary recurrence | 24 months
  Axillary recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence in lymph nodes draining the primary tumour site, i.e. nodes in the ipsilateral axilla, infraclavicular fossa, supraclavicular fossa and interpectoral area. The date of axillary recurrence is the date on which imaging or pathology report (whichever comes first) confirms axillary recurrence.
Axillary recurrence | 36 months
  Axillary recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence in lymph nodes draining the primary tumour site, i.e. nodes in the ipsilateral axilla, infraclavicular fossa, supraclavicular fossa and interpectoral area. The date of axillary recurrence is the date on which imaging or pathology report (whichever comes first) confirms axillary recurrence.
Axillary recurrence | 48 months
  Axillary recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence in lymph nodes draining the primary tumour site, i.e. nodes in the ipsilateral axilla, infraclavicular fossa, supraclavicular fossa and interpectoral area. The date of axillary recurrence is the date on which imaging or pathology report (whichever comes first) confirms axillary recurrence.
Axillary recurrence | 60 months
  Axillary recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence in lymph nodes draining the primary tumour site, i.e. nodes in the ipsilateral axilla, infraclavicular fossa, supraclavicular fossa and interpectoral area. The date of axillary recurrence is the date on which imaging or pathology report (whichever comes first) confirms axillary recurrence.
Regional (nodal) recurrence | 12 months
  Regional (nodal) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrent tumour in the lymph nodes in the ipsilateral axilla, infraclavicular, supraclavicular fossa, interpectoral area or ipsilateral internal mammary chain. The date of regional recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Regional (nodal) recurrence | 24 months
  Regional (nodal) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrent tumour in the lymph nodes in the ipsilateral axilla, infraclavicular, supraclavicular fossa, interpectoral area or ipsilateral internal mammary chain. The date of regional recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Regional (nodal) recurrence | 36 months
  Regional (nodal) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrent tumour in the lymph nodes in the ipsilateral axilla, infraclavicular, supraclavicular fossa, interpectoral area or ipsilateral internal mammary chain. The date of regional recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Regional (nodal) recurrence | 48 months
  Regional (nodal) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrent tumour in the lymph nodes in the ipsilateral axilla, infraclavicular, supraclavicular fossa, interpectoral area or ipsilateral internal mammary chain. The date of regional recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Regional (nodal) recurrence | 60 months
  Regional (nodal) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrent tumour in the lymph nodes in the ipsilateral axilla, infraclavicular, supraclavicular fossa, interpectoral area or ipsilateral internal mammary chain. The date of regional recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Disease free survival | 12 months
  Disease-Free Survival (DFS); defined and calculated as the time from targeted sentinel node biopsy until the date of first event of either a loco-regional invasive breast cancer relapse, distant relapse, ipsilateral or contralateral new invasive primary breast cancer or death by any cause or the censor date.
Disease free survival | 24 months
  Disease-Free Survival (DFS); defined and calculated as the time from targeted sentinel node biopsy until the date of first event of either a loco-regional invasive breast cancer relapse, distant relapse, ipsilateral or contralateral new invasive primary breast cancer or death by any cause or the censor date.
Disease free survival | 36 months
  Disease-Free Survival (DFS); defined and calculated as the time from targeted sentinel node biopsy until the date of first event of either a loco-regional invasive breast cancer relapse, distant relapse, ipsilateral or contralateral new invasive primary breast cancer or death by any cause or the censor date.
Disease free survival | 48 months
  Disease-Free Survival (DFS); defined and calculated as the time from targeted sentinel node biopsy until the date of first event of either a loco-regional invasive breast cancer relapse, distant relapse, ipsilateral or contralateral new invasive primary breast cancer or death by any cause or the censor date.
Disease free survival | 60 months
  Disease-Free Survival (DFS); defined and calculated as the time from targeted sentinel node biopsy until the date of first event of either a loco-regional invasive breast cancer relapse, distant relapse, ipsilateral or contralateral new invasive primary breast cancer or death by any cause or the censor date.
Overall survival | 12 months
  Overall survival; calculated as the time from targeted sentinel node biopsy until the date of death by any cause or the censor date.
Overall survival | 24 months
  Overall survival; calculated as the time from targeted sentinel node biopsy until the date of death by any cause or the censor date.
Overall survival | 36 months
  Overall survival; calculated as the time from targeted sentinel node biopsy until the date of death by any cause or the censor date.
Overall survival | 48 months
  Overall survival; calculated as the time from targeted sentinel node biopsy until the date of death by any cause or the censor date.
Overall survival | 60 months
  Overall survival; calculated as the time from targeted sentinel node biopsy until the date of death by any cause or the censor date.
Local (breast or chest wall) recurrence | 12 months
  Local (breast or chest wall) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence after mastectomy in the skin or soft tissue of the chest wall within the anatomical area bounded by the mid-sternal line, the clavicle, the posterior axillary line and the costal margin or any type of breast carcinoma in the breast after conservation therapy. The date of local recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Local (breast or chest wall) recurrence | 24 months
  Local (breast or chest wall) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence after mastectomy in the skin or soft tissue of the chest wall within the anatomical area bounded by the mid-sternal line, the clavicle, the posterior axillary line and the costal margin or any type of breast carcinoma in the breast after conservation therapy. The date of local recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Local (breast or chest wall) recurrence | 36 months
  Local (breast or chest wall) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence after mastectomy in the skin or soft tissue of the chest wall within the anatomical area bounded by the mid-sternal line, the clavicle, the posterior axillary line and the costal margin or any type of breast carcinoma in the breast after conservation therapy. The date of local recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Local (breast or chest wall) recurrence | 48 months
  Local (breast or chest wall) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence after mastectomy in the skin or soft tissue of the chest wall within the anatomical area bounded by the mid-sternal line, the clavicle, the posterior axillary line and the costal margin or any type of breast carcinoma in the breast after conservation therapy. The date of local recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.
Local (breast or chest wall) recurrence | 60 months
  Local (breast or chest wall) recurrence is defined as pathologically (cytology or biopsy) and/or radiologically confirmed recurrence after mastectomy in the skin or soft tissue of the chest wall within the anatomical area bounded by the mid-sternal line, the clavicle, the posterior axillary line and the costal margin or any type of breast carcinoma in the breast after conservation therapy. The date of local recurrence is the date on which the imaging or pathology report (whichever comes first) confirms local recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Goyal, Study Chair — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (10):
- United Kingdom (10):
  - Burnley General Teaching Hospital, Burnley
  - Addenbrooke's Hospital, Cambridge
  - University Hospitals of Derby and Burton, Derby
  - Gartnavel General Hospital, Glasgow
  - Wycombe Hospital, High Wycombe
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Royal Alexandra Hospital, Paisley
  - The Shrewsbury and Telford Hospital NHS Trust, Shrewsbury
  - Mersey and West Lancashire Teaching Hospitals, St Helens
  - The Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No